CLINICAL TRIAL: NCT07293221
Title: Use of Immersive Virtual Reality for the Management of Anxiety Among Nurses : a Randomized Trial
Brief Title: Immersive Virtual Reality for the Management of Anxiety Among Nurses
Acronym: RVI-Nurse
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SCP Anesthésie - Réanimation de la Clinique du Pont de Chaume (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RVI-Nurse
Record Dates: First submitted 2025-09-22; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Anxiety; Nurse Based Care Management
Keywords: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: nurses will be randomized into two parallel, open-label groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hypnotic Immersive Virtual Reality Group (Active Comparator): * On the day of the study, upon arrival in the coffee break room, nurses complete the Spielberger self-assessment anxiety questionnaire.
  * The anesthesiologist responsible for the protocol (Dr. PEREIRA DE SOUZA) ensures that the nurse has understood the study protocol and answers any questions.
  * The nurse then begins the hypnotic immersive VR session in a calm, dedicated room.
  * At the end of the session, before returning to work, the nurse completes the Spielberger questionnaire again, along with a Likert scale to evaluate satisfaction. Any potential adverse effects (nausea, vomiting, etc.) are also recorded.
  Interventions: Other: virtual reality
- Control Group (No Intervention): * On the day of the study, upon arrival in the coffee break room, nurses complete the Spielberger questionnaire.
  * The anesthesiologist (Dr. PEREIRA DE SOUZA) ensures understanding of the protocol and answers questions.
  * The nurse then takes their coffee break normally with their team.
  * At the end of the coffee break, before returning to work, the nurse completes the Spielberger questionnaire again, along with the Likert scale.

INTERVENTIONS:
Other: virtual reality — Since 2024, the investigators have offered hypnotic VR sessions to nurses at the Clinique du Pont de Chaume to better manage their anxiety. Despite the high satisfaction rate reported in our questionnaires, the investigators now aim to statistically evaluate the efficacy of this intervention. Ultimately, these results could justify a broader investment in this type of equipment, making it available to a larger number of healthcare professionals (orderlies, nursing assistants, secretaries, pharmacists, physicians, etc.), but only if this complementary intervention demonstrates scientific efficacy.
  Arms: Hypnotic Immersive Virtual Reality Group

SUMMARY:
The nursing profession is recognized as one of the most demanding in the healthcare sector. Constant exposure to illness, suffering, and death, combined with an increasing workload, leads to fatigue, stress, and especially persistent anxiety. This anxiety affects not only the psychological and physical health of nurses but also the quality of care provided. From an organizational perspective, anxiety promotes absenteeism, demotivation, and turnover, creating a vicious cycle of collective exhaustion.

To relieve their anxiety, an increasing number of healthcare providers are turning to complementary medicine, particularly immersive virtual reality (VR) interventions.

Immersive VR hypnosis has been used for several years as a non-pharmacological approach to anxiety management. It constitutes a relational experience engaging both physiological and psychological mechanisms, allowing the user to improve their experience and reduce or even eliminate anxiety.

Randomized clinical trials conducted in recent years have evaluated the efficacy of immersive VR hypnosis. Some results indicate that it reduces anxiety more significantly than pharmacological treatments in control groups and is at least as effective as other complementary therapies (relaxation, massage, acupuncture, yoga, etc.). However, the strength of these conclusions remains limited due to a substantial risk of methodological bias. Rigorous new studies, with strict control conditions, are required, particularly regarding the efficacy of hypnosis applied to nurses.

Since 2024, the investigators have offered hypnotic VR sessions to nurses at the Clinique du Pont de Chaume to better manage their anxiety. Despite the high satisfaction rate reported in our questionnaires, the investigators now aim to statistically evaluate the efficacy of this intervention. Ultimately, these results could justify a broader investment in this type of equipment, making it available to a larger number of healthcare professionals but only if this complementary intervention demonstrates scientific efficacy.

DETAILED DESCRIPTION:
Research Hypothesis The hypothesis of this study is that hypnotic immersive virtual reality (VR) interventions can reduce nurses' anxiety.

Benefit/Risk Assessment The use of hypnotic immersive VR techniques presents no risk to nurses. This approach is complementary to existing protocols, notably by providing immersive VR headsets during rest periods.

________________________________________ Research Objectives Primary Objective To evaluate the efficacy of hypnotic immersive VR in reducing anxiety among day-shift nurses before and after a coffee break.

Secondary Objective To assess the effect of hypnotic immersive VR on nurses' satisfaction following the coffee break.

Study Design This is a pilot, open-label, randomized controlled trial (RCT), conducted intention-to-treat, single-center, aiming to evaluate the efficacy of hypnotic immersive virtual reality (VR) interventions on day-shift nurses' anxiety after a coffee break.

The protocol is initially limited to day-shift nurses for organizational reasons and to maintain group homogeneity. Night-shift nurses are exposed to different constraints: smaller staff, altered circadian rhythm, limited number of physicians, etc.

The secondary objective of this study is to assess the impact of this intervention on nurses' satisfaction.

________________________________________ Study Endpoints Primary Endpoint The primary endpoint is the change in the Spielberger anxiety score, measured between the beginning and the end of the coffee break.

Secondary Endpoint The secondary endpoint is the nurses' satisfaction, measured using a Likert scale.

________________________________________ Study Timeline Start of recruitment: Upon obtaining all regulatory approvals. Recruitment period: 24 months. Duration of participation per nurse: 1 day (maximum delay between inclusion and data collection).

Total study duration: 27 months. Pre-Inclusion and Inclusion Visits Pre-inclusion visit: Conducted by Dr. PEREIRA DE SOUZA NETO 2 weeks to 1 month before data collection. During this visit, the nurse is informed about the protocol, its objectives, constraints, potential risks (nausea, vomiting), and expected benefits. A copy of the information sheet and consent form is provided for reflection.

Inclusion visit: Conducted by Dr. PEREIRA DE SOUZA on the day of data collection. The nurse provides written informed consent. Both the nurse and investigator sign and date the consent form. Copies are distributed as follows:

One copy is given to the nurse. The original is kept by Dr. PEREIRA DE SOUZA in a secure location inaccessible to third parties, even in case of staff reassignments during the study.

ELIGIBILITY:
Inclusion Criteria:

Nurses who have received appropriate information, agreed to participate, and signed the informed consent form.

Nurses working day shifts (06:00-18:00) with a coffee break scheduled from 09:00 to 09:15.

Exclusion Criteria:

Nurses who have not provided informed consent or cannot comply with the study protocol.

History of photosensitive epilepsy or seizures. Unstable vestibular disorders or a severe history of motion sickness preventing the use of immersive VR.

Employer refusal if participation cannot be organized outside work obligations (participation must remain voluntary and without professional consequences).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in the Spielberger questionnaire measurement | From enrollement to the end of study at 1 day
  To evaluate the efficacy of hypnotic immersive VR in reducing anxiety among day-shift nurses before and after a coffee break. Anxiety will be measured with the Spielberger anxiety score, measured between the beginning and the end of hypnotic immersive VR or between the beginning and the end of the coffee break or

SECONDARY OUTCOMES:
The secondary endpoint is the nurses' satisfaction, measured using a Likert scale. | From enrollement to the end of study at 1 day
  At the end of the session, before returning to work, the nurse completes the Likert scale to evaluate satisfaction. Any potential adverse effects (nausea, vomiting, etc.) are also recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Edmundo P PEREIRA DE SOUZA NETO, Phd, Principal Investigator — Clinique du Pont de Chaume - Montauban

IPD SHARING:
Plan to Share IPD: Yes
Data collection is performed by Dr. PEREIRA DE SOUZA NETO, and data management by a Data Manager of the Clinical Research and Innovation Department of Clinique du Pont de Chaume.
  Any transfer of all or part of the study database is decided by the sponsor and formalized in a written agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At the end of the study
Access Criteria: All information required by the protocol must be recorded in the electronic patient record.
  Study Monitoring
  * Logistics and monitoring:
    * Managed by the Clinical Research Associate (CRA) in collaboration with the principal investigator.
    * Includes organizing inclusions, participant follow-up, and protocol compliance control.
  * Progress reports:
    * The CRA prepares and submits regular progress reports to the sponsor.
    * Reports include recruitment, adverse events, and collected data.

REFERENCES:
- [Background] Williamson A. What is hypnosis and how might it work? Palliat Care. 2019 Jan 31;12:1178224219826581. doi: 10.1177/1178224219826581. eCollection 2019. No abstract available. PMID 30728719
- [Background] Vaughn F, Wichowski H, Bosworth G. Does preoperative anxiety level predict postoperative pain? AORN J. 2007 Mar;85(3):589-604. doi: 10.1016/S0001-2092(07)60130-6. PMID 17352896
- [Background] Tefikow S, Barth J, Maichrowitz S, Beelmann A, Strauss B, Rosendahl J. Efficacy of hypnosis in adults undergoing surgery or medical procedures: a meta-analysis of randomized controlled trials. Clin Psychol Rev. 2013 Jul;33(5):623-36. doi: 10.1016/j.cpr.2013.03.005. Epub 2013 Mar 26. PMID 23628907
- [Background] Spielberger CD. State-Trait Anxiety Inventory for adults sampler set manual, instrument and scoring guide. Mind Garden Eds. 1983, 1-75.
- [Background] Sharar SR, Miller W, Teeley A, Soltani M, Hoffman HG, Jensen MP, Patterson DR. Applications of virtual reality for pain management in burn-injured patients. Expert Rev Neurother. 2008 Nov;8(11):1667-74. doi: 10.1586/14737175.8.11.1667. PMID 18986237
- [Background] Pozek JJ, De Ruyter M, Khan TW. Comprehensive Acute Pain Management in the Perioperative Surgical Home. Anesthesiol Clin. 2018 Jun;36(2):295-307. doi: 10.1016/j.anclin.2018.01.007. Epub 2018 Apr 7. PMID 29759289
- [Background] Noergaard MW, Hakonsen SJ, Bjerrum M, Pedersen PU. The effectiveness of hypnotic analgesia in the management of procedural pain in minimally invasive procedures: A systematic review and meta-analysis. J Clin Nurs. 2019 Dec;28(23-24):4207-4224. doi: 10.1111/jocn.15025. Epub 2019 Sep 3. PMID 31410922
- [Background] Mavros MN, Athanasiou S, Gkegkes ID, Polyzos KA, Peppas G, Falagas ME. Do psychological variables affect early surgical recovery? PLoS One. 2011;6(5):e20306. doi: 10.1371/journal.pone.0020306. Epub 2011 May 25. PMID 21633506
- [Background] Madden K, Middleton P, Cyna AM, Matthewson M, Jones L. Hypnosis for pain management during labour and childbirth. Cochrane Database Syst Rev. 2012 Nov 14;11:CD009356. doi: 10.1002/14651858.CD009356.pub2. PMID 23152275
- [Background] Kendrick C, Sliwinski J, Yu Y, Johnson A, Fisher W, Kekecs Z, Elkins G. Hypnosis for Acute Procedural Pain: A Critical Review. Int J Clin Exp Hypn. 2016;64(1):75-115. doi: 10.1080/00207144.2015.1099405. PMID 26599994
- [Background] Ip HY, Abrishami A, Peng PW, Wong J, Chung F. Predictors of postoperative pain and analgesic consumption: a qualitative systematic review. Anesthesiology. 2009 Sep;111(3):657-77. doi: 10.1097/ALN.0b013e3181aae87a. PMID 19672167
- [Background] Flory N, Salazar GM, Lang EV. Hypnosis for acute distress management during medical procedures. Int J Clin Exp Hypn. 2007 Jul;55(3):303-17. doi: 10.1080/00207140701338670. PMID 17558720
- [Background] Fisch S, Brinkhaus B, Teut M. Hypnosis in patients with perceived stress - a systematic review. BMC Complement Altern Med. 2017 Jun 19;17(1):323. doi: 10.1186/s12906-017-1806-0. PMID 28629342
- [Background] Facco E, Casiglia E, Masiero S, Tikhonoff V, Giacomello M, Zanette G. Effects of hypnotic focused analgesia on dental pain threshold. Int J Clin Exp Hypn. 2011 Oct-Dec;59(4):454-68. doi: 10.1080/00207144.2011.594749. PMID 21867380
- [Background] Elkins GR, Barabasz AF, Council JR, Spiegel D. Advancing Research and Practice: The Revised APA Division 30 Definition of Hypnosis. Am J Clin Hypn. 2015 Apr;57(4):378-85. doi: 10.1080/00029157.2015.1011465. PMID 25928776
- [Background] Chan PY, Scharf S. Virtual Reality as an Adjunctive Nonpharmacological Sedative During Orthopedic Surgery Under Regional Anesthesia: A Pilot and Feasibility Study. Anesth Analg. 2017 Oct;125(4):1200-1202. doi: 10.1213/ANE.0000000000002169. PMID 28598921
- [Background] Berliere M, Roelants F, Watremez C, Docquier MA, Piette N, Lamerant S, Megevand V, Van Maanen A, Piette P, Gerday A, Duhoux FP. The advantages of hypnosis intervention on breast cancer surgery and adjuvant therapy. Breast. 2018 Feb;37:114-118. doi: 10.1016/j.breast.2017.10.017. Epub 2017 Nov 11. PMID 29136523
- [Background] Benhaiem JM, Attal N, Chauvin M, Brasseur L, Bouhassira D. Local and remote effects of hypnotic suggestions of analgesia. Pain. 2001 Jan;89(2-3):167-73. doi: 10.1016/s0304-3959(00)00359-6. PMID 11166472
- [Background] Askay SW, Patterson DR, Sharar SR. VIRTUAL REALITY HYPNOSIS. Contemp Hypn. 2009 Mar;26(1):40-47. doi: 10.1002/ch.371. PMID 20737029